CLINICAL TRIAL: NCT04996654
Title: Feasibility, Usability and Acceptance of a Newly Developed Exergame-Based Traininng Concept for Older Adults With Mild Neurocognitive Disorder - A Pilot Randomized Controlled Trial
Brief Title: Feasibility of a Novel Exergame-Based Training Concept for Older Adults With Mild Neurocognitive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eling DeBruin (Other)
Responsible Party: Sponsor-Investigator, Eling DeBruin, Prof. Dr., Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EK 2021-N-79
Record Dates: First submitted 2021-07-11; First posted 2021-08-09 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Mild Neurocognitive Disorder
Keywords: Exergames; Mild Neurocognitive Disorder; Cognition; Feasibility; Usability
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: Allocation ration = 2 (Exergame Group) : 1 (Usual Care)
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluator of the pre- and post-measurements will be blinded to group allocation. For all data assessed throughout the intervention period (i.e. only applicable for the intervention group), blinding of investigators is not possible. Blinding of participants was also not possible since usual care will be used as a control intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame (Experimental): Participants will perform a twelve-week training intervention in addition to their usual care as provided by the memory clinics where the patients are recruited. The training intervention will be prescribed according to a newly developed exergame-based intervention concept that consists of an individually adapted multi-domain exergame-based simultaneous cognitive-motor training with incorporated cognitive tasks that will be adopted with a deficit-oriented focus on the neurocognitive domains of (1) learning and memory, (2) executive function, (3) complex attention, and (4) perceptual-motor function.
  Interventions: Behavioral: Exergame
- Usual Care (Active Comparator): An active control group will proceed with usual care as provided by the memory clinics where the patients are recruited.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Exergame — According to the training concept, each participant is instructed to train 5x/week for 21 min per session resulting in a weekly exercise volume of 105 min. All training sessions are planned to take place at participant's homes using the exergame training system Dividat Senso (Dividat AG, Schindellegi, Switzerland; CE certification).
  Arms: Exergame
Behavioral: Usual Care — An active control group will proceed with usual care as provided by the memory clinics where the patients are recruited.
  Arms: Usual Care

SUMMARY:
The primary objective of this pilot study is to evaluate the feasibility (i.e. recruitment, adherence, compliance, attrition), usability (i.e. system usability), and acceptance (i.e. enjoyment, training motivation and perceived usefulness) of a newly developed exergame-based intervention concept for older adults with mNCD. As a secondary objective, preliminary effects of the intervention on cognition, brain resting-state functional connectivity, gait, cardiac autonomic regulation, and psychosocial factors (i.e. quality of life, and levels of depression, anxiety, and stress) will be explored. This allows to synthesize data for a sample size calculation on basis of a formal power calculation for a future RCT.

A two-arm, parallel-group, single-blinded (i.e. outcome evaluator of pre- and post-measurements blinded to group allocation) pilot randomized controlled study with an allocation ration of 2 : 1 (i.e. intervention : control) including 17 - 25 older adults with mNCD will be conducted between June and December 2021. The active control group will proceed with usual care as provided by the memory clinics where the patients are recruited. The intervention group will perform a twelve-week training intervention according to a newly developed exergame-based intervention concept in addition to usual care. Primary outcomes will be assessed throughout the training intervention period. The measurements of all secondary outcomes will be conducted at ETH Hönggerberg within two weeks prior to starting (PRE) and after completing (POST) the study intervention.

DETAILED DESCRIPTION:
After recruitment, interested subjects will be screened on eligibility between July and September 2021. All potential subjects will be fully informed about the study procedures by providing verbal explanations and an information sheet. Expected effects, benefits and risks of the study will be explained by the investigator, who will also be available to answer open questions and clarify uncertainties of participants. It will further be verified, that withdrawal is permitted at any time during the study without giving any reason. After sufficient time for considerations, suitable patients willing to take part in the study will provide written informed consent prior to any measurements and the first study appointment will be scheduled. At the first scheduled appointment, pre-measurements (PRE) will be performed. Thereafter, participants will be randomly allocated to the intervention group (i.e. 'exergame group') or active control group (i.e. 'usual care'). Subsequently, participants in the exergame group will be familiarized with the exergame training system 'Dividat Senso' (Dividat AG, Schindellegi, Switzerland; CE certification), and the study intervention will be started according to the newly developed exergame-based intervention concept. After completing the twelve-week training intervention, post-measurements (POST) will be performed for both groups. Both, the pre- and the post-measurements will take place and within two weeks prior to starting or after completing the intervention.

INTERVENTIONS:

Usual Care:

An active control group will proceed with usual care as provided by the memory clinics where the patients are recruited.

Exergame Group:

Participants will perform a twelve-week training intervention in addition to their usual care as provided by the memory clinics where the patients are recruited. The training intervention will be prescribed according to a newly developed exergame-based intervention concept. The training intervention concept was planned and reported using the Consensus on Exercise Reporting Template (CERT): It consists of an individually adapted multi-domain exergame-based simultaneous cognitive-motor training with incorporated cognitive tasks that will be adopted with a deficit-oriented focus on the neurocognitive domains of (1) learning and memory, (2) executive function, (3) complex attention, and (4) perceptual-motor function. According to the training concept, each participant is instructed to train 5x/week for 21 min per session resulting in a weekly exercise volume of 105 min. All training sessions are planned to take place at participant's homes using the exergame training system Dividat Senso (Dividat AG, Schindellegi, Switzerland; CE certification). In case the training cannot be performed at home, the training sessions will be performed at ETH Hönggerberg and the instructed training frequency is reduced to 3x/week for 21 min per session resulting in a weekly volume of 63 min. Nonetheless, it is still recommended to train at the suggested optimal frequency (5x/week) and volume (105 min/week).

The training concepts is structured in three phases. It starts with a familiarization period of two weeks. During this phase, most of the training sessions (i.e. 4 out of 5 sessions) are supervised. After this initial guided familiarization period, supervision of training sessions is gradually reduced to 1x/week during a four-week transition phase. This transition phase aims to lead participants to being able to train independently. In this transition phase, the amount of supervision of training sessions is individually determined within a predefined range in accordance with the capabilities and preferences of the participants. From the 7th week until completion of the training intervention, semi-autonomous training with one supervised training session per week are prescribed for each participant.

Throughout the training intervention period, all sessions will be prescribed following the same basic structure: Each session consists of three blocks with 3 phases per block. Phase 1 - Facilitation aims to apply a moderate physical intensity in the context of challenging but feasible cognitive and motoric demands mainly intending to trigger neurophysiological mechanisms, which promote neuroplasticity while additionally using cognitive stimulation to guide these neuroplastic processes. This phase includes games focusing on neurocognitive domains that are least impaired. The external task demand is individually adapted to ensure an appropriate internal training load. More specifically, the internal training load is subdivided into a fixed component (i.e. physical intensity) and a variable component (i.e. neurocognitive (game-) demand). An additional stepping task is used to set the level of physical intensity. It includes walking on the spot at a predefined stepping frequency that is needed to reach a moderate level of physical intensity (i.e. ranging between 40 and 59 % heart rate reserve (HRR))). The stepping frequency will be individually determined for each participant. A battery figure add-on is visible in the center of the screen that provides real-time visual feedback whether the predefined stepping frequency is reached. More specifically, if the predefined minimal required stepping frequency is reached or exceeded, the battery stays at equilibrium or fills. As long as the battery level is above 80 % (indicated by a line), the battery stays green. If the participants' stepping frequency falls below the predefined minimal required stepping frequency, the battery level decreases, and the battery turns orange (40 - 80 %) or red (below 40 %) indicating that the stepping frequency should be increased. On top of this fixed physical intensity, a variable amount of neurocognitive (game-) demands (e.g. game type, task complexity, predictability of required tasks) is applied. Since the physical intensity is kept constant, changes in the overall internal training load can mainly be attributed to these neurocognitive and motoric (game-) demands and, accordingly, the internal training load can be adjusted on basis of these game characteristics. Therefore, the neurocognitive demands of the exergame are individually adapted in order to ensure an appropriate total internal training load. The monitoring and adaption of the internal training load will be based on predefined progression rules for adapting characteristics of external training load. Phase 2 - Guidance aims to make use of the triggered neurophysiological mechanisms from phase 1 to specifically guide neuroplastic processes of the mainly impaired neurocognitive domain. Therefore, games focusing on the mainly impaired neurocognitive domain for the individual participant (e.g. amnestic single domain => learning and memory) are used. These games solely focus on cognitive and motoric demands, but not on physical exercise intensity. The cognitive-motoric demands of the exergame (also called 'external load') are individually adapted in order to ensure an appropriate internal training load. The monitoring and adaption of the internal training load will be based on predefined progression rules for adapting characteristics of external training load. Phase 3 - Coherence aims to implement a structured approach as a surrogate for the breaks between games. More specifically, resonance breathing training guided by heart rate variability biofeedback (HRVB) is used. HRVB training is a behavioral intervention aiming to increase cardiac autonomic control, to enhance homeostatic regulation, and to regulate emotional state. It includes paced breathing for two minutes following the rhythm of the individually predetermined resonance frequency visualized on the screen of the exergame device. The resonance frequency will be evaluated for each participant before starting the training intervention.

ELIGIBILITY:
Inclusion Criteria:

* (Group 1 = mNCD) clinical diagnosis of 'Mild Neurocognitive Disorder' (mNCD) according to the International Classification of Diseases 11th Revision (ICD-XI) OR (Group 2 = sMCI) patients screened for mild cognitive impairment (sMCI) according to the following criteria: (a) informant (i.e. healthcare professionals)-based suspicion of MCI confirmed by (b) an objective screening of MCI based on the German Version of the Quick Mild Cognitive Impairment Screen with (b1) a recommended cut-off score for cognitive impairment (MCI or dementia) of < 62/100, while (b2) not falling below the cut-off score for dementia (i.e. < 45/100), while (c) activities of daily living remain intact.
* fully vaccinated against coronavirus (SARS-CoV-2) with a Federal Office of Public Health (FOPH)-approved mRNA vaccine
* German speaking
* age ≥ 50 years
* able to stand at least for 10 min without assistance

Exclusion Criteria:

* mobility impairments (i.e. gait, balance) that prevent experiment participation
* presence of additional neurological disorders (i.e. epilepsy, stroke, multiple sclerosis, Parkinson's disease, brain tumors, or traumatic disorders of the nervous system)
* presence of any other unstable or uncontrolled diseases
* additional Covid-19 specific exclusion criteria (according to the Federal Office of Public Health):

  * high blood pressure (self-reported; systolic ≥ 140 mmHg and/or Diastolic ≥ 90 mmHg)
  * Chronic respiratory condition
  * Diabetes
  * Condition or therapy that weakens the immune system
  * Cardiovascular Disease
  * Cancer (present and/or under treatment)
  * Serious obesity (BMI ≥ 40 kg/m2)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Feasibility - recruitment (relative) | Through recruitment completion, an average of 12 weeks.
  recruitment rate (relative) [%] = number of screened people / number of enrolled participants
Feasibility - recruitment (absolute) | Through recruitment completion, an average of 12 weeks.
  recruitment rate (absolute) [] = number of eligible participants recruited per month
Feasibility - adherence | Through recruitment completion, an average of 12 weeks.
  adherence rate [%] = total number of training sessions attended / total number of training sessions offered
Feasibility - compliance | Through recruitment completion, an average of 12 weeks.
  compliance rate [%] = total training duration attended [min] / total training duration offered [min]
Feasibility - attrition | Through recruitment completion, an average of 12 weeks.
  attrition rate = number of drop-outs / number of enrolled participants
Usability | System Usability is assessed in the Exergame Group at week 6 of the study intervention.
  Usability will be assessed on basis of the validated German version of the System Usability Scale (SUS-DE). The SUS-DE is assessed in week 6 of the exergame-based intervention. It consists of ten items that are rated on a five-point Likert scale (i.e. ranging from 1 - "strongly disagree" to 5 - "strongly agree"). A total score will be calculated according to the scoring guidelines of the SUS. The total SUS score ranges between 0 and 100, whereas higher scores indicate better usability. A total SUS score of at least 70 will be considered an "acceptable" solution (i.e. 52 = ok, 73 = good, 85 = excellent, 100 = best imaginable).
Acceptance - enjoyment | Through recruitment completion, an average of 12 weeks.
  Enjoyment of the exergame-based intervention concept will be assessed on basis of the Exergame Enjoyment Questionnaire (EEQ) that will be translated to German according to the guidelines for the process of cross-cultural adaptation of self-report measures. It consists of 20 statements corresponding to four categories of questions: (1) immersion, (2) intrinsically rewarding activity, (3) control, and (4) exercise. Each statement will be responded to on a five-point Likert scale (i.e. strongly disagree (1 point), disagree (2 points), neutral (3 points), agree (4 points), and strongly agree (5 points). The EEQ will be analyzed by calculating the average overall score as well as an average score for each category of questions.
Acceptance - motivation | Through recruitment completion, an average of 12 weeks.
  The quality (of type) and quantity (of level) of training motivation will be assessed using of the German version of the Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3) that is a widely used, valid and reliable measure of the continuum of motivation for exercise in different areas. It consists of 24 items assessing behavioral regulation in exercise contexts on a 5- point Likert scale ranging from 0 = 'not true for me' to 4 = 'very true for me'.
Acceptance - perceived usefulness | Through recruitment completion, an average of 12 weeks.
  Perceived usefulness will be evaluated on basis of patient-interviews, organized as semi-structured interviews along a predefined interview guide.

SECONDARY OUTCOMES:
Changes in Global Cognition | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  The German Version of the Quick Mild Cognitive Impairment Screen (Qmci) will be used to assess the overall level of cognitive functioning of the study population. The Qmci can be completed within 3 - 5 minutes and is scored as a point rate out of a maximum score of 100. It comprises six subtests: orientation (10 points), registration (5 points), clock drawing (15 points), delayed recall (20 points), verbal fluency (20 points), and logical memory (30 points). The recommended cut-off score for cognitive impairment (MCI or dementia) is < 62/100. The Qmci will be administered according to its guidelines.
Changes in Learning and Memory - Part 1 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Learning and memory will be assessed using the German version of the subtests 'logical memory' of the Wechsler Memory Scale-Revised (WMS-R-LM). The WMS-IV-LM is a measure of auditory verbal contextual learning and memory and has demonstrated excellent reliability and validity. The validated German version of the WMS-IV-LM will be used. Two short stories (Story A and B) will be read aloud to the participant. The participant will be instructed to recall details of the stories immediately (WMS-IV-LM I, immediate recall) and after a delay of 30 min (WMS-IV-LM II, delayed recall). The Older Adults battery (for ages 65 or older) will be used for all participants. The test will be instructed and conducted according to the standardized administration and scoring manual. During the 30 minutes retention phase, unrelated assessment (e.g. gait analysis) will be performed that to not interfere with memory.
Changes in Learning and Memory - Part 2 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Learning and memory will be assessed using a computerized version of the Digit Span Forward test (PEBL Digit Span Forward (PEBL-DSF)). The PEBL-DSF test will be used to assess immediate recall, short-term attention span and information processing speed. It will be executed using the PEBL Test battery software (Version 2.1 (2)). Participants will have to remember and repeat digit sequences that will be presented on the screen in the correct order. Span length will cover two to eight digits. For each digit span, two trials will be presented to the participant prior to increasing sequence length. For every correct replication of a digit sequence, one point will be scored, summing up to a total point score. Additionally, the length of the longest correctly repeated digit sequence will be recorded as the maximum span. Instructions will be presented on the screen and will be explained verbally to each participant before starting the task.
Changes in Complex Attention - Part 1 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Complex attention will be assessed using a computerized version of the Trail Making Test - Part A (PEBL-TMT-A). The TMT-A is valid and reliable neuropsychological tests to assess psychomotor processing speed and visuoperceptual abilities. It consists of 25 randomly allocated circles distributed over a sheet of paper. Participants will be asked to connect encircled numbers in ascending order. A computerized version of the of the TMT-A (PEBL Test battery software (Version 2.1 (2)) will be used in this study since it provides more precise measurements. The test will be explained and demonstrated prior to starting the test procedure and a short practice session will be conducted. Participants will be instructed to perform the test as quickly as possible. Completion time will be limited to 300 seconds. Completion times [s] (including the time for correction of errors) and number of errors will be measured.
Changes in Complex Attention - Part 2 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Complex attention will be assessed using the subtests 'Alertness' of the Test of Attentional Performance (TAP Alertness). The TAP Alertness was designed to determine intrinsic and phasic attention under two conditions. The first condition (A) requires participants to react to a cross appearing at randomly varying intervals on the screen by pressing a switch as fast as possible. In the second task (B), responses will only be required when preceded by a warning tone. 20 target stimuli will be presented for each condition in the order 'ABBA' to compensate for the effects of fatigue. Reaction times will be measured. Median reaction times reflect general reaction speed attenuation, while the variability of reaction times indicates the stability of performance, that is, the consistency with which attention is focused.
Changes in Complex Attention - Part 3 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Complex attention will be assessed using the subtests 'Go-NoGo' of the Test of Attentional Performance (TAP Go-NoGo). The TAP Go-NoGo will be used to assess selective attention and inhibition. Two different stimuli will be presented on the screen alternating in sequence representing test form '1 of 2'. Participants' task will be to react as quickly as possible to the appearance of the diagonal cross (x) by pushing the button and suppress their reaction to appearing upright crosses (+).
Changes in Executive Function - Part 1 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  To measure planning ability, the HOTAP-A will be used. A set of photo cards containing actions typical for everyday life (e.g. making coffee, washing clothes, shopping) will be presented. The requirement consists in the correct sorting of photo cards on which individual sub-steps of typical everyday actions (e.g. making coffee, doing the laundry, shopping) are depicted. Every correctly rearranged picture will be granted one point. The outcome variable will be the sum of the points divided by the time they needed to arrange the cards. The test will be administered according to the protocol of the manufacturer.
Changes in Executive Function - Part 2 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  The PEBL Digit Span Backward (PEBL-DSB) test will be used to assess working memory capacity. It will be executed using the PEBL Test battery software (Version 2.1 (2)). Participants will have to remember and repeat digit sequences that will be presented on the screen in reverse order. Span length will cover two to eight digits. For each digit span, two trials will be presented to the participant prior to increasing sequence length. For every correct replication of a digit sequence, one point will be scored, summing up to a total point score. Additionally, the length of the longest correctly repeated digit sequence will be recorded as the maximum span. Instructions will be presented on the screen and will be explained verbally to each participant before starting the task.
Changes in Executive Function - Part 3 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Cognitive inhibition will be assessed using the subtests 'Incompatibility' of the Test of Attentional Performance (TAP Incompatibility).
Changes in Executive Function - Part 4 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Complex attention will be assessed using a computerized version of the Trail Making Test - Part B (PEBL-TMT-B). It consists of 25 randomly allocated circles distributed over a sheet of paper. In the TMT-B, circles include numbers (1 - 13) and letters (A - L) which will need to be connected in ascending order alternated between numbers and letters (i.e. 1 - A - 2 - B - 3 - C, etc.).
Changes in Perceptual-Motor Function | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Visuo-spatial functions will be tested with a computerized version of the classic Shepard and Metzler's mental rotation task. The PEBL Mental Rotation Task (PEBL MRT) will be executed using the PEBL Test battery software (Version 2.1 (2)). Instructions will be presented on the screen and will be explained verbally to each participant before starting the task. Pairs of differently rotated two-dimensional polygons will be presented simultaneously on the screen. Participants will need to decide as quickly as possible whether the two presented objects are identical (i.e. pressing <Lshift> on the keyboard) or different (i.e. pressing <Rshift> on the keyboard). Reaction times [s] as well as performance (number of correct answered trials) will be measured. The measured reaction times of correct answered trials of the PEBL MRT will serve as an indicator for mental rotation ability.
Changes in Brain Functional Connectivity | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Surface EEG activity will be recorded at a sampling frequency of 1000 Hz by a high-density 64-channel EEG system (eego sport, ANT Neuro, Enschede, The Netherlands). Three EEG cap sizes will be employed in order to accommodate different head circumferences and EEG electrodes will be placed according the 10-10 international system. EEG reference and ground will be placed over the left and right mastoid, respectively. An electrodes impedance ≤ 10 kΩ will be required before EEG recordings. The measurement will be conducted at the same conditions as the measurement of resting heart rate and HRV including twice 2 mins with eyes opened (focussing on a visual cue), 2 mins eyes closed. Resting EEG data will be analyzed with connectivity analysis (i.e. functional connectivity in the delta-theta band as a robust signature of conscious states).
Changes in Spatiotemporal Gait Parameters | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor. The BTW G-sensor will be attached with semi-elastic belt to the lower back (i.e. at the height of the second lumbar spinal process below the imaginary line connecting the left and right most prominent bone of the posterior superior iliac spine) of the participant. A validated gait-analysis protocol consisting of a figure-8 walking path (i.e. distance approximately 7 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability (i.e. cadence, gait speed, stride duration, stride length, stance phase duration, swing phase duration, double support time, and single support time). Therefore, participants will perform ten repetitions of the figure-8 walking path during at preferred walking speed.
Changes in vagally-mediated Heart Rate Variability (HRV) | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  To determine changes in resting HRV, all participants will be instructed to sit in a comfortable position on a chair without speaking, both feet flat on the floor with knees at a 90° angle, hands on thighs, and eyes closed. The measurement (10 min acclimatization followed by 5 min resting measurement) will be performed in a quiet room with dimmed light and at room temperature, using the heart rate monitor (Polar M430) and sensor (Polar H10). Mainly vagal-mediated HRV indices (i.e. mean R-R time interval (mRR), root mean square of successive RR interval differences (RMSSD), the percentage of successive RR intervals that differ by more than 50 ms (pNN50), the absolute power of the high-frequency band, the relative power of HF (in normal units), the Poincaré plot standard deviation perpendicular to the line of identity (SD1), and the parasympathetic nervous system tone index (PNS-Index) will be calculated using Kubios HRV Premium.
Changes in Psychosocial Factors - Part 1 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Quality of life will be evaluated in interview format using the Quality of Life-Alzheimer's Disease (QOL-AD) scale. The QOL-AD is a valid and reliable self-report 13-item scale assessing various domains of QOL of cognitively impaired patients including "patient's physical condition, mood, interpersonal relation-ships, ability to participate in meaningful activities, financial situation, and an overall assessment of self as a whole and quality of life as a whole". Comparable values for patients with mNCD are available. Each item is rated on a 4-point Likert scale (i.e. "poor" (1 point), "fair" (2 point), "neutral" (3 points), and "excellent" (4 points)). The overall score will be computed by summing the scores of the 13 items, resulting in an overall score ranging between 13 and 52, whereas higher scores indicating higher QOL. The German version of the QOL-AD scale will be used.
Changes in Psychosocial Factors - Part 2 | Both, the pre- and the post-measurements of secondary outcome measurements will take place and within two weeks prior to starting or after completing the intervention.
  Levels of depression, anxiety, and stress will be assessed using the short version of the Depression, Anxiety and Stress Scale-21 (DASS-21). It is a self-report questionnaire consisting of 21 items including seven questions for each of the three indicators (i.e. depression, anxiety and stress). Each item contains a statement that is rated on a four-point Likert scale (i.e. "did not apply to me at all" (0 points), "applied to me to some degree, or some of the time" (1 point), "applied to me to a considerable degree, or a good part of time" (2 points), and "applied to me very much, or most of the time" (3 points)) regarding the extent to which the statement applied within the previous week. Scores for each indicator will be calculated by summing the scores for the corresponding items multiplied by two. The resulting scores range between 0 and 42, whereas higher scores indicate higher levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Eling D de Bruin, PhD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Result] Manser P, Poikonen H, de Bruin ED. Feasibility, usability, and acceptance of "Brain-IT"-A newly developed exergame-based training concept for the secondary prevention of mild neurocognitive disorder: a pilot randomized controlled trial. Front Aging Neurosci. 2023 Sep 21;15:1163388. doi: 10.3389/fnagi.2023.1163388. eCollection 2023. PMID 37810620